CLINICAL TRIAL: NCT04177849
Title: Örebro Multicenter Study on Operative Treatment of Cervical Radiculopathy: Anterior Cervical Decompression and Fusion Versus Posterior Foraminotomy
Brief Title: Örebro Multicenter Study on Operative Treatment of Cervical Radiculopathy
Acronym: OMSAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Örebro County (Other)
Collaborators: Uppsala University Hospital (Other); Rygglkirurgiskt Centrum Stockholm AB (Other); Norrlands University Hospital (Other)
Responsible Party: Principal Investigator, Marek Holy, Principal Investigator, Head of Spine Unit, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-00003
Record Dates: First submitted 2019-11-19; First posted 2019-11-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cervical Radiculopathy; Cervical Root Compression
Keywords: Pain; Nerve root dysfunction; Anterior Cervical Decompression and Fusion; Posterior Foraminotomy
MeSH Terms: conditions — Radiculopathy; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior Cervical Decompression and Fusion (ACDF) (Active Comparator): Patients entered into this arm are treated via an anterior approach with disk excision, root canal decompression and fusion of the affected segment with a cage and plate.
  Interventions: Procedure: ACDF
- Posterior Foraminotomy (PF) (Experimental): Patients entered into this arm are treated via a posterior approach through intermuscular planes. The root canal is decompressed by burring the medial third of the facet joint. No fusion is performed.
  Interventions: Procedure: PF

INTERVENTIONS:
Procedure: ACDF — A 4-cm anterolateral transverse incision is made over the index level, on either the right or left side. Platysma is sectioned transversal to its fibers and the anterior aspect of the spinal column is bluntly exposed between the carotid sheath and the esophagus. The disk is excised, including the posterior longitudinal ligament. Disk fragments and/or osteophytes from the uncovertebral joint on the affected side are removed until the root is fully decompressed. Reconstruction is typically done with an interbody spacer, autologous bone graft and a stabilizing plate screwed to the adjacent vertebral bodies. A fusion cage with integrated screws may also be used according to the surgeon's preference.
  Arms: Anterior Cervical Decompression and Fusion (ACDF)
Procedure: PF — A 4-cm longitudinal midline incision exposes the spinous processes of the adjacent vertebrae. The facet joint covering the index foramen is exposed through intermuscular planes. The root canal is opened as the medial third of the facet joint is removed with a high-speed diamond burr. The affected nerve root is decompressed by laterally undercutting the facet joint throughout its length.
  Arms: Posterior Foraminotomy (PF)

SUMMARY:
This study compares anterior cervical decompression and fusion (ACDF) to posterior foraminotomy (PF) in surgical treatment for cervical radiculopathy (CR) caused by root canal compression, in a multicenter prospective randomized trial. The investigators hypothesize equal decompression of nerve root, and equal clinical outcome in both treatment groups.

DETAILED DESCRIPTION:
Both ACDF and PF are effective in surgical treatment of CR. However, the techniques has different complication profiles and carry different costs. No comparative study with high level of evidence has been published, why the basis for clinical guidelines are lacking.

The study consists of 110 patients with CR not responding to non-surgical treatment for 6 weeks and with a Neck Disability Index (NDI) over 30 points/60 %, that are randomized to either technique in a 1:1 ratio and followed for two years.

Primary variable is NDI, secondary variables are Numerical Pain Rating Scale (NRS) separately for arm and neck pain and health related quality of life (EQ-5D). Tertiary variables are complications and reoperations. The patients are also followed radiographically with plain x-rays in extension and flexion, CT, and MRI.

The study has a non-inferiority design with ACDF as active control. A NDI difference of less than 8,5 points/17 % (=minimally clinical important difference, MCID, for NDI) is considered a non-inferior result. A secondary superiority evaluation will also be performed.

Analysis Primarily, patient-related outcome measures will be analyzed in terms of intention to treat (ITT) and include all randomized patients. Missing values will be imputed. The investigators will calculate, by using analysis of covariance (ANCOVA), the mean outcome values for each treatment group, adjusted for baseline values of the outcome. The mean difference between the groups will also be presented.

Secondary outcome analyses using the Student t test, Chi-Square, Mann-Whitney, Fisher exact test.

The tertiary outcome analyses will be based on available cases. The time to revision surgery according to treatment assignment will be analyzed and plotted according to the Kaplan-Meier method, while hazard ratios, with regard to having secondary surgery after ACDF compared to PF, will be estimated by the Cox model with calendar time as the time scale. Men and women will be analyzed separately.

An "Ad Interim" analysis will be performed by a non-partial observer and/or statistician when 40 patients are included, regarding NDI difference, complications and reoperations.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of radiating arm pain with duration of at least six weeks
* Neck disability index (NDI) over 30 points (60%);
* Correlating findings on MRI on one or two cervical levels
* Eligible for both treatments
* Ability to understand and read Swedish.

Exclusion Criteria:

* Previous cervical spine surgery
* More then two cervical levels requiring treatment
* Severe facet joint osteoarthritis
* Symptoms or marked radiologic signs of myelopathy
* Drug abuse
* Dementia or expected low compliance
* Cervical malformation
* Marked instability, 3.5-mm translation or >11 degrees more motion compared to adjacent segments
* History of severe cervical trauma
* Generalized pain syndrome or WAD
* Pregnancy
* Rheumatoid arthritis
* Ankylosing spondylitis
* Malignancy
* Active infection or another severe systemic disease
* Patients that are unsuitable for either intervention deemed by the consultant spine surgeon

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Neck Disability index, NDI. | 4-6 weeks, 3 months, 1 year, 2 year, 5 year
  Primary variable is NDI change at two year compared to baseline. NDI is a self-administered questionnaire with 10 items measuring disability in patients with neck pain. The questions cover daily activities, such as the ability to dress, lift heavy objects, read, work, drive a car, sleep and perform leisure time activities, as well as the amount of pain, headache and concentration abilities. Each item is scored from 0 to 5. MCID for NDI is 7,5-8,5 or 17,3%.
  NDI change will also be measured at different time intervals to highlight the change over time.

SECONDARY OUTCOMES:
EQ-5D | 4-6 weeks, 3 months, 1 year, 2 year, 5 year
  Secondary variable is EQ-5D change at two year compared to baseline. EQ-5D, The European Quality of Life-5 Dimensions (EQ-5D; with a range from approximately -0.5 to 1, with higher scores indicating better quality of life) using the Swedish translation [36, 37].
  EQ-5D change will also be measured at different time intervals to highlight the change over time.
NRS neck, NRS arm | 4-6 weeks, 3 months, 1 year, 2 year, 5 year
  Numerical Rating Scale (NRS) for pain is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number 0 no pain to 10 worst pain imaginable that best reflects the intensity of their pain. MCID is 2.2 point for NRS
  NRS change will also be measured at different time intervals to highlight the change over time

CONTACTS AND LOCATIONS:
Overall Officials: Per Wretenberg, Prof. MD. PhD, Study Chair — Region Örebro County; Claes Olerud, Prof. MD. PhD, Study Director — Uppsala University
Locations (4):
- Sweden (4):
  - Universistessjukhuset Örebro, Örebro
  - Ryggkirurgiskt Centrum Stockholm, Stockholm
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska Sjukhuset Uppsala, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holy M, MacDowall A, Sigmundsson FG, Olerud C. Operative treatment of cervical radiculopathy: anterior cervical decompression and fusion compared with posterior foraminotomy: study protocol for a randomized controlled trial. Trials. 2021 Sep 8;22(1):607. doi: 10.1186/s13063-021-05492-2. PMID 34496941